CLINICAL TRIAL: NCT04711577
Title: Examining Self-tracking Behaviors in a Mobile Intervention for Binge Eating and Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Andrea Graham, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00213531
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Binge Eating
MeSH Terms: conditions — Obesity; Bulimia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1 (Experimental): Track clinician-determined symptoms
  Interventions: Behavioral: Track clinician-determined symptoms
- Condition 2 (Experimental): Track clinician-determined and self-determined symptoms
  Interventions: Behavioral: Track clinician-determined and self-determined symptoms

INTERVENTIONS:
Behavioral: Track clinician-determined symptoms — Participants will track clinician-determined symptoms
  Arms: Condition 1
Behavioral: Track clinician-determined and self-determined symptoms — Participants will track clinician-determined symptoms and a self-determined symptom
  Arms: Condition 2

SUMMARY:
The purpose of this study is to understand users' experiences and interests completing self-tracking in a mobile intervention for binge eating and weight management.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Obesity (BMI ≥30)
* Recurrent binge eating (≥12 episodes in the past 3 months)
* Interested in losing weight and reducing binge eating
* Willing to use a mobile application
* Willing to practice self-monitoring
* Has access to a scale
* Not pregnant
* English-speaking

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Compliance | 3 weeks
  Number of tracking entries completed
Satisfaction with tracking | 3 weeks
  Self-reported satisfaction with tracking, based on the Satisfaction subscale of the Usefulness, Satisfaction, and Ease of use (USE) Questionnaire, with higher scores on the 1-7 rating scale indicating greater satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States